CLINICAL TRIAL: NCT02380144
Title: Bioavailability of Carotenoids and Flavonoids From Fresh Oranges and Orange Juice.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Hohenheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: F-2013-097
Record Dates: First submitted 2015-02-23; First posted 2015-03-05 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: carotenoid; bioavailability; beta-cryptoxanthin; flavonoid; hesperidin; narirutin; randomized cross-over; Pharmacokinetics; micronutrients; Oranges/Orange Juice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orange Fruit - Orange Juice (Experimental): Sequence of test foods during the intervention period:
  1st: Orange fruit; 2nd: Orange juice
  Interventions: Other: Fresh orange fruit and pasteurized fruit juice
- Orange Juice - Orange Fruit (Experimental): Sequence of test foods during the intervention period:
  1st: Orange juice; 2nd: Orange fruit
  Interventions: Other: Fresh orange fruit and pasteurized fruit juice

INTERVENTIONS:
Other: Fresh orange fruit and pasteurized fruit juice

SUMMARY:
The study was designed as a randomized 2-way cross-over study to assess the bioavailability of carotenoids and flavonoids from sweet oranges and orange juice. Volunteers followed a wash-out period for 2 weeks prior to eating either 400 g of fresh oranges or 719 g of orange juice. The amount of test food was adjusted to deliver an equal amount of β-cryptoxanthin (740 µg). After a consecutive wash-out period of 2 weeks, the procedure was repeated and the volunteers ingested the complementary test food. Blood samples were collected at 8 time points up to 9.5 h after test meal consumption. Additionally, 24 h-urine was collected to evaluate flavonoid recovery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women
* BMI: 17-60
* Age: 18-65

Exclusion Criteria:

* Women who are lactating or pregnant or plan to be pregnant
* Individuals using tobacco products
* Individuals with metabolic or malabsorption disorders
* Individuals with a history of cancer
* Individuals with a history of liver insufficiency
* Individuals with a history of chronic and lipid metabolism-related diseases
* Individuals with an allergy to oranges
* Obese individuals (BMI > 30)

Ages: 23 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Mean AUC (nmol/L*9.5 h) of beta-cryptoxanthin concentration in blood plasma chylomicrons after ingestion of fresh oranges and orange juice, respectively. | 0 - 9.5 h after each intervention

SECONDARY OUTCOMES:
Mean AUC of hesperidin- and narirutin-metabolite concentration in blood plasma after ingestion of fresh oranges and orange juice, respectively. | 0 - 9.5 h after each intervention
Mean hesperetin and naringenin concentration (µmol/L) in 24 h-urine after ingestion of fresh oranges and orange juice, respectively. | 0 - 24 h after each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Reinhold Carle, Prof. Dr., Principal Investigator — University of Hohenheim
Locations (1):
- Chair of Plant Foodstuff Technology and Analysis (150d), University of Hohenheim, Stuttgart, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] Aschoff JK, Rolke CL, Breusing N, Bosy-Westphal A, Hogel J, Carle R, Schweiggert RM. Bioavailability of beta-cryptoxanthin is greater from pasteurized orange juice than from fresh oranges - a randomized cross-over study. Mol Nutr Food Res. 2015 Oct;59(10):1896-904. doi: 10.1002/mnfr.201500327. Epub 2015 Jul 20. PMID 26114420